CLINICAL TRIAL: NCT07352826
Title: The Effect of Blood Carboxyhemoglobin Levels on NF-kB, NRF2 and PGC-1α During Low-flow and Normal-flow Anesthesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Veysel Koksal, MD, Principal Investigator, Ataturk Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: B.30.2.YYU.0.01.00.00/91
Record Dates: First submitted 2025-09-15; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Anesthesia
Keywords: low flow anesthesia; COHb; NF-kB; NRF2; PGC-1 alpha

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- COHb (Experimental)
  Interventions: Behavioral: low-flow anasthesia; Behavioral: Normal akımlı anestezi
- TAS (Experimental)
  Interventions: Behavioral: low-flow anasthesia; Behavioral: Normal akımlı anestezi
- TOS (Experimental)
  Interventions: Behavioral: low-flow anasthesia; Behavioral: Normal akımlı anestezi
- HIF 1a (Experimental)
  Interventions: Behavioral: low-flow anasthesia; Behavioral: Normal akımlı anestezi

INTERVENTIONS:
Behavioral: low-flow anasthesia — In Group LF, FGF will then be maintained at 0.6 L/min (O₂ 50%, air 50%), with desflurane adjusted to maintain MAC = 1
Behavioral: Normal akımlı anestezi — In Group NF, FGF will be maintained at 2 L/min (O₂ 50%, air 50%) with desflurane adjusted to maintain MAC = 1..

SUMMARY:
Carbon monoxide (CO) is a colorless, odorless, and tasteless gas that exerts diverse biological effects across tissues and organs. At high concentrations, it is recognized as toxic because of harmful effects such as tissue hypoxia, oxidative stress, peroxynitrite formation, inflammation, apoptosis, and immune damage. However, the endogenous production of CO suggests that it may confer protective mechanisms to the host. These protective effects include inhibition of platelet activation, smooth muscle relaxation, vasoactive properties, anti-inflammatory and anti-apoptotic actions, and beneficial influences on neurotransmission. Despite its toxic potential, low-concentration endogenous CO may provide protection linked to the body's defense mechanisms. In this study, we aimed to investigate the anti-apoptotic effects of carbon monoxide at low concentrations. To this end, the relationships between COHb levels and plasma levels of NF-κB, NRF2, and PGC-1α were analyzed statistically.

DETAILED DESCRIPTION:
A total of 120 patients aged 18-70 years, classified as ASA I and scheduled for inhalational anesthesia lasting ≥2 hours, will be included. Patients with cardiovascular disease, respiratory system disease, hepatic or renal disease; pregnant or breastfeeding women; trauma patients; those undergoing emergency surgery; procedures lasting <2 hours; those receiving intraoperative blood transfusion; smokers; and individuals who decline participation will be excluded.

All participants who agree to join the study will read and sign an informed consent form describing the study. Preoperative evaluations will be performed 1 day before surgery. Thirty minutes before surgery, a 22G intravenous cannula will be inserted, and 8 mL of blood will be drawn into a yellow-cap gel biochemistry tube and 1.5 mL into a blood gas syringe containing 60 IU of dry heparin. Biochemistry samples will be centrifuged at 4000 rpm for 10 minutes in the medical biochemistry laboratory. The separated sera will be transferred to Eppendorf tubes and stored at -80 °C until the day of analysis. Blood gas samples will be analyzed on a blood gas analyzer (Radiometer ABL 520, Copenhagen, Denmark). After blood sampling, an infusion of 0.9% sodium chloride (NaCl) at 10 mL/kg/h will be initiated. Patients will receive IV premedication with 1.5 mg midazolam; on the operating table, ECG, noninvasive blood pressure, and peripheral oxygen saturation (SpO₂) will be monitored. Before induction, all patients will undergo preoxygenation with O₂ at 6 L/min via face mask for 3 minutes.

For induction of anesthesia, fentanyl 1 µg/kg (Fentanyl Citrate, Abbott Laboratories, North Chicago, USA) and propofol 2 mg/kg IV (Propofol, Fresenius Kabi, Sweden) will be administered over 20-30 seconds. After loss of the eyelash reflex, rocuronium bromide 0.6 mg/kg (Esmeron, Organon, Netherlands) will be given IV for neuromuscular blockade, and endotracheal intubation will be performed with a cuffed tube of appropriate size for the patient's age and body habitus. Following propofol administration and until intubation, all patients will be manually ventilated with 100% O₂. After intubation, mechanical ventilation will be provided with an anesthesia machine (Datex-Ohmeda Aisys CS2, Madison, USA) in volume-controlled mode with a tidal volume of 6-8 mL/kg, respiratory rate of 12-14/min, and PEEP of 5 cmH₂O. Soda lime will be used as the CO₂ absorbent (Sorbolime, Berkim, Türkiye), and replacement of the absorbent will be verified before induction for each patient.

Patients will be randomly assigned to one of two groups: Group LF (low-flow, n=60) and Group NF (normal-flow, n=60). In both groups, fresh gas flow (FGF) will be set at 4 L/min (O₂ 50%, air 50%) until the minimum alveolar concentration (MAC) reaches 1. In Group LF, FGF will then be maintained at 0.6 L/min (O₂ 50%, air 50%), with desflurane adjusted to maintain MAC = 1. In Group NF, FGF will be maintained at 2 L/min (O₂ 50%, air 50%), with desflurane adjusted to maintain MAC = 1. In both groups, blood sampling will be repeated at the 2nd hour of surgery.

During the final 30 minutes of surgery, patients will receive postoperative analgesia consisting of tramadol HCl (Contramal, Türkiye) 100 mg IV, paracetamol (Partemol, Türkiye) 1 g IV, and dexketoprofen (Ketavel, Türkiye) 50 mg IV. In the normal-flow group, after placement of the final skin suture, the inhalational agent will be discontinued and the carrier gas switched to 100% O₂; FGF will be increased to 8 L/min. In the low-flow group, the inhalational agent will be discontinued 20 minutes before the anticipated end of surgery; FGF will be maintained at 0.6 L/min until the final skin suture and then increased to 8 L/min. After the return of spontaneous breathing, neostigmine 0.03 mg/kg (Plantigmin, Türkiye) and atropine 0.01 mg/kg (Turktıpsan, Türkiye) will be administered in both groups to achieve extubation.

Postoperatively, patients will be transferred to the post-anesthesia care unit, where respiratory and hemodynamic parameters will be monitored for 30 minutes before transfer to the ward. In both groups, blood sampling will be repeated at postoperative hour 24 using the same method. The following variables will be recorded: duration of anesthesia, SpO₂, venous blood gas results, hemodynamic parameters, postoperative recovery time and quality, and postoperative complications (e.g., nausea and vomiting). Blood samples obtained in the preoperative, intraoperative, and postoperative periods will be centrifuged and stored at -80 °C. Following biochemical analysis, COHb, NF-κB, NRF2, and PGC-1α levels will be subjected to statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

aged 18-70 years

classified as ASA I

scheduled for inhalational anesthesia lasting ≥2 hours

Exclusion Criteria:

Patients with cardiovascular disease, respiratory system disease, hepatic or renal disease

pregnant or breastfeeding women

trauma patients

those undergoing emergency surgery

procedures lasting <2 hours

those receiving intraoperative blood transfusion

smokers

individuals who decline participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Blood COHb, NF-kB, NRF2, and PGC-1α levels during Low-Flow and Normal-Flow Anesthesia | 24 HOUR
  COHb concentrations
Blood COHb, NF-kB, NRF2, and PGC-1α levels during Low-Flow and Normal-Flow Anesthesia | 24 HOUR
  NF-kB concentrations
Blood COHb, NF-kB, NRF2, and PGC-1α levels during Low-Flow and Normal-Flow Anesthesi | 24 HOUR
  NRF2 concentrations
Blood COHb, NF-kB, NRF2, and PGC-1α levels during Low-Flow and Normal-Flow Anesthesi | 24 HOUR
  PGC-1α concentrations

CONTACTS AND LOCATIONS:
Locations (1):
- Veysel, Erzurum, Turkey (Türkiye)